CLINICAL TRIAL: NCT05730972
Title: Transcutaneous Electrical Acupoint Stimulation (TEAS) for the Treatment of Pain in Bone Metastases of Lung Cancer: A Multicenter Prospective RCT Study
Brief Title: TEAS for the Treatment of Pain in Bone Metastases of Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Yi Liang, Professor, Chief Chinese Medicine Practitioner, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021ZZ017; 2021ZZ017 (Other Grant/Funding Number: the Key Foundation of Chinese Medicine Research Program of Zhejiang Province); 2014KYA162 (Other Grant/Funding Number: General Research Plan of Medicine and Health of Zhejiang Province)
Record Dates: First submitted 2023-01-28; First posted 2023-02-16 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cancer Pain; Non Small Cell Lung Cancer; Bone Metastases; Acupuncture
Keywords: transcutaneous electrical nerve stimulation; Transcutaneous electrical acupoint stimulation
MeSH Terms: conditions — Cancer Pain; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- true TEAS (Experimental): A pair of conductive gel patch, connecting to the Huatuo SDZ-ⅡB portable electronic needle therapy instrument, are respectively affixed to the ipsilateral Jiaji acupoint group (EX-B2) or the ipsilateral limb acupoint group(Hegu (LI4) - Waiguan (TE5), or Zusanli (ST36) - Sanyinjiao (SP6)), so as contralateral side.
  A single TEAS treatment takes 30 min. TEAS specific parameters were dilatation wave 2Hz and stimulus current intensity in degrees as tolerated by the patient.
  7 days was considered as 1 session. Self-controlled treatment refers to not setting an upper limit on the number of treatment times, but must have met at least 3 days or 5 times of TEAS treatment within each session.
  A total of 4 sessions of treatment were administered.
  Interventions: Device: Transcutaneous electrical acupoint stimulation; Drug: Routine palliative treatment
- sham TEAS (Sham Comparator): Each step of the sham TEAS operation is the same as the TEAS group. A total of 4 sessions of treatment were administered. 10 free TEAS treatments will be given after the trial.
  Interventions: Device: Sham transcutaneous electrical acupoint stimulation; Drug: Routine palliative treatment

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — The patients are taken in the recumbent or sitting position, and the local skin at the acupoints is routinely disinfected. A pair of conductive gel patch, connecting to the Huatuo SDZ-ⅡB portable electronic needle therapy instrument, are respectively affixed to the ipsilateral acupoint group, so as contralateral side.
  Other Names: TEAS
  Arms: true TEAS
Device: Sham transcutaneous electrical acupoint stimulation — The electroacupuncture instrument has a normal screen display as the Huatuo SDZ-ⅡB portable electronic needle therapy instrument, but could not output current normally.
  Other Names: sham TEAS
  Arms: sham TEAS
Drug: Routine palliative treatment — The patients in both groups received routine palliative treatment of tumors, such as chemotherapy, immunotherapy, targeted therapy, drug analgesic therapy, nutrition support, and so on.

SUMMARY:
This multicenter, prospective, randomized controlled research study aims to objectively evaluate the role of transcutaneous electrical acupoint stimulation (TEAS), which combines the theory of acupuncture with transcutaneous electrical nerve stimulation (TENS) therapy, for the treatment of pain in patients with bone metastases from lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the diagnostic criteria of non-small cell lung cancer and had a diagnosis of definite bone-metastatic-related pain.
* Potent opioid analgesics have been prescribed regularly.
* Bone protective agents (bisphosphonates or desumumab) have been used regularly.
* Expected survival ≥ 3 months with no obvious contraindication to opioid therapy.
* Stable vital signs and ECOG-PS score ≤ 2 points; able to cooperate with researchers to complete relevant study evaluations.
* Signed informed consent.

Exclusion Criteria:

* Definitively diagnosed with pain unrelated to lung cancer.
* Received local radiation therapy or surgery targeting bone metastases within 1 week before enrollment or will receive during the intervention period. The surgery including vertebroplasty, radioparticle implantation, neurological lesions, and other minimally invasive interventions.
* Venous thrombosis in the upper and lower extremities (below the elbow / knee joint), active cerebrovascular disease, severe cardiopulmonary dysfunction, or those with respiratory depression.
* Pacemaker implantation or metallic implants in vivo.
* Skin lesions at the acupoints, poor skin condition, or other situations that are not suitable for treatment with TEAS.
* Opioid hypersensitivity.
* Psychiatric disorders or severe cognitive deficits.
* Participating in other clinical trialists influencing the evaluation of the results of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The response rate of average pain in the brief pain inventory (BPI) at the end of week 4 | week 4
  According to the international consensus on palliative radiotherapy endpoints for bone metastasis clinical trials, the degree of therapeutic response for bone metastatic pain can be classified as complete response (CR: pain score of 0 and no increase in daily oral morphine equivalent dose (OMED) ), partial response (PR: ①pain score decrease of ≥ 2 and no increase in OMED; ②pain score no increase and decrease of ≥ 25% in OMED), pain progression (PP: ①≥ 2 increase in pain score with no decrease in OMED; ②≥ 1 increase in pain score with ≥ 25% increase in OMED) and indeterminate response (IR: cases not classified as CR / PR / PP).
  Subjects in which complete or partial relief of pain was achieved were pain responders; Subjects whose pain progressed or was indeterminate response were non responders. The response rate of average pain = ((CR+PR) / No. of subjects) *100%.

SECONDARY OUTCOMES:
The changes of pain and inference scores in Brief Pain Inventory | week 4, week 8, week 12
The changes of frequency of breakthrough pain within 1 week | week 4, week 8, week 12
The changes of OMED on assessment days | week 4, week 8, week 12
  The daily oral morphine equivalent dose over the past 24 h will be recorded for both groups at each testing time point. Equivalent morphine dose conversions will be established in accordance with the NCCN clinical practice guidelines for adult cancer pain (version 3.2022). For instance, fentanyl transdermal patch (25 mcg/h) will be considered approximately equal to oxycodone (30 mg/d), parenteral morphine (20 mg/d), and oral morphine (60 mg/d).
Quality of life measured by EORTC QLQ-C30 score | week 4, week 8, week 12
  The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) is an integrated system for assessing the quality of life (QoL) of cancer patients. The EORTC QLQ-C30 incorporates nine multi-item scales: five functional scales (Physical, Role, Cognitive, Emotional and Social Functioning); three symptom scales (Fatigue, Pain and Nausea/Vomiting); and a Global Health Status/QoL scale. Six single item scales are also included (Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties). Scale scores were calculated by averaging items within scales and transforming average scores linearly. All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
The changes in mood scale scores of Hamilton Rating Scale for Depression (HAM-D) | week 4, week 8, week 12
  HAM-D is a standardized scale for the measurement of the severity of depressive symptoms, initially designed to yield a total score based on 17 items. The scores of anxiety/depression and its change during the previous 2 weeks from baseline will be recorded.The total score > 24 points, severe depression. 17≤ score ≤24, moderate depression. 7≤ score ≤17, mild depression. < 7 points, no depressive symptoms.
The changes in mood scale scores of Hamilton Rating Scale for Hamilton Rating Scale for Anxiety (HAM-A) | week 4, week 8, week 12
  HAM-A is one of the most widely used rating scales to measure the severity of perceived anxiety symptoms. A total of 14 items were included 14 items. The total score ≥29 points, may be severe anxiety. ≥21 points, there must be obvious anxiety. ≥14 points, must have anxiety. ≥7 points, may have anxiety. < 7 points, no anxiety symptoms.
The changes of tri-lineage cell counts in blood | week 4, week 8, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Yi Liang, PhD, Study Chair — Zhejiang Chinese Medical University, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyu Z, Shen Q, Tian S, Gong L, Lou H, Bao G, Wu Z, Lu C, Zhang W, Huang R, Ji C, Zheng S, Pan W, Ying Y, Jin J, Liang Y. Effects of Patient-Controlled Transcutaneous Electrical Acupoint Stimulation on Cancer Induced Bone Pain Relief in Patients with Non-Small Cell Lung Cancer: Study Protocol for a Randomized Controlled Trial. J Pain Res. 2024 Mar 26;17:1285-1298. doi: 10.2147/JPR.S437296. eCollection 2024. PMID 38560406